CLINICAL TRIAL: NCT04018677
Title: TOGETHER: Track Outcomes and Guidance, Technology for Health and Effective Resources
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Medable Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-44783; VAR0182 (Other: OnCore); IRB-44783 (Other: Stanford IRB)
Record Dates: First submitted 2019-06-18; First posted 2019-07-12 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beta Testing (Experimental): For the beta testing, input will be provided by cancer patient/survivor, caregivers, and clinicians. TOGETHER app will be downloaded on smart phone. Subjects will be asked to answer questions and/or perform activities on his/her smartphone device. Project information will include responses to surveys and giving additional feedback on app user experience.
  Interventions: Behavioral: Use of TOGETHERCare app
- Usability testing (Experimental): For the usability testing, caregivers will be the primary type of stakeholder providing input. TOGETHER app will be downloaded on smart phone. Subjects will be asked to answer questions and/or perform activities on his/her smartphone device. Project information will include responses to surveys and giving additional feedback on app user experience.
  Interventions: Behavioral: Use of TOGETHERCare app

INTERVENTIONS:
Behavioral: Use of TOGETHERCare app — TOGETHERCare (Medable Inc.) is a mobile software application on a smart software system that informal caregivers can use to develop and implement home-based care for cancer patients/survivors. It is intended to improve the care experience by helping to alleviate the cancer care-giving burden and facilitate communication with patients' healthcare teams by centering the conversation around a care plan.

SUMMARY:
The goal of this project is to iteratively develop and test a TOGETHER pilot mobile app product in preparation for commercialization. TOGETHER is a mobile application on a smart software system that informal caregivers can use to develop and implement home-based care for cancer patients/survivors.

The Technical Objectives are to:

1. Establish the project team and obtain stakeholder feedback on what to include in the product.
2. Evaluate IT customization requirements and HIPAA compliance security, and privacy protocols.
3. Develop a prototype to show NCI and then a pilot version for beta and usability testing among stakeholders.
4. Enhance interoperability and test integration into health system(s) - if feasible.
5. Develop user support documentation for stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18 years or older) who are either:

  * Cancer patient/survivor receiving care or with plans to transition to care in the community setting.
  * Caregiver of cancer patient/survivor receiving care or with plans to transition to care in the community setting.
  * Clinician of cancer patient/survivor receiving care or with plans to transition to care in the community setting.
* Cancer patient is a patient of Stanford Health Care.
* Patient, Caregiver, and Clinician are willing to be connected on the app.
* Have a smartphone and data plan that allows for app installation and usage.
* Must speak, read and write in English, because all study materials and communication will be in English.

Exclusion Criteria:

* Patient does not have a cancer diagnosis.
* Cancer patient/survivor is not receiving care or does not have plans to transition to care in the community setting.
* Cancer patient is not a patient of Stanford Health Care.
* Patient, Caregiver, and Clinician are not willing to be connected on the app.
* Unable to speak, read and write in English.
* Does not have a smartphone nor data plan that allows for app installation and usage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Assess user experience with TOGETHER app | 1 year
  User experiences will be assessed by measuring overall experiences.
Assess user experience with TOGETHER app | 1 year
  User experiences will be assessed by measuring module recommendation.
Assess user experience with TOGETHER app | 1 year
  User experiences will be assessed by measuring dynamics/flow of app use, module recommendation, and general demographics.
Assess user experience with TOGETHER app | 1 year
  User experiences will be assessed by measuring problems with app use.
Assess caregiver's experience with TOGETHER app | 1 year
  Caregiver's experience with TOGETHER app will be assessed for clarity of documentation.
User documentation feedback | 1 year
  General feedback/recommendations for the app, including user documentation feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Vasu Divi, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oakley-Girvan I, Davis SW, Kurian A, Rosas LG, Daniels J, Palesh OG, Mesia RJ, Kamal AH, Longmire M, Divi V. Development of a Mobile Health App (TOGETHERCare) to Reduce Cancer Care Partner Burden: Product Design Study. JMIR Form Res. 2021 Aug 13;5(8):e22608. doi: 10.2196/22608. PMID 34398787